CLINICAL TRIAL: NCT07201831
Title: ACT on MASH: A Multi-country, Cross-sectional Quantitative Study Exploring Awareness, Understanding, and Perceptions of the Relation Between Cardiorenal Metabolic Conditions and MASLD/MASH Among Healthcare Providers, People With MASLD/MASH, and At-risk Population
Brief Title: A Multi-country, Cross-sectional Quantitative Study Exploring Awareness, Understanding, and Perceptions of the Relation Between Cardiorenal Metabolic Conditions and MASLD/MASH Among Healthcare Providers, People With MASLD/MASH, and At-risk Population
Acronym: MASH
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-8185; U1111-1308-2796 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-09-18; First posted 2025-10-01 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Dysfunction-associated Steatohepatitis (MASH)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCP Group: This group includes Health Care Practitioners (HCPs) who self-report to being at least somewhat familiar with Metabolic dysfunction-associated steatohepatitis (MASH)
  Interventions: Other: No treatment given
- Patient Groups: This group includes patients diagnosed with Metabolic dysfunction-associated steatohepatitis (MASH), diagnosed with Metabolic Associated Steatotic Liver Disease (MASLD), or at risk for development/diagnosis of MASH
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this study is to collect information for scientific research and to better understand awareness and to understand overall risk awareness, diagnoses and treatment related to liver related diseases. The study aims to collect valid responses through online questionnaires from the participants. This study is a survey-based study without collection of laboratory data. It will take the participant 25 minutes to complete the survey. The study is not related to any specific treatment options or pharmaceutical product.

ELIGIBILITY:
Inclusion Criteria:

HCP inclusion criteria

* Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Licensed to practice medicine in one of the countries of interest: United States, Canada, France, Germany, Japan
* Must be a practicing endocrinologist, hepatologist, cardiologist, obesity specialist, primary care physician, radiologist, nurse practitioner or physician assistant (NP/PA US only)
* Must be at least "somewhat familiar" (as opposed to "not at all familiar) with Metabolic dysfunction-associated steatohepatitis (MASH) (do not need to be currently treating people with MASH) 6. Must have at least 2 years in practice 7. Must spend at least 50 percentage of their time in patient care

Diagnosed patient inclusion criteria

* Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Diagnosis of MASH or Metabolic Associated Steatotic Liver Disease (MASLD) within past 24 months
* Live in one of the countries of interest: United States, Canada, France, Germany, Japan
* Have at least one comorbid condition: obesity, pre-diabetes, type 2 diabetes (T2D), metabolic syndrome, dyslipidaemia, hypertension, cardiovascular disease, chronic kidney disease

At risk patient inclusion criteria

* Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* Male or female, age above or equal to 18 years at the time of signing informed consent.
* Live in one of the countries of interest: United States, Canada, France, Germany, Japan
* Must have one or more risk factors associated with MASH [obesity, pre-diabetes, type 2 diabetes (T2D), metabolic syndrome, dyslipidaemia, hypertension, cardiovascular disease, chronic kidney disease], be diagnosed with steatosis (incidental finding) or have a blood test that shows raised liver enzymes.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes two population segments. The first segment is made up of Health Care Practitioners (HCPs) who self-report to being at least somewhat familiar with Metabolic dysfunction-associated steatohepatitis (MASH). The second segment consists of three subsegments defined as people who have been diagnosed with MASH, or people who have been diagnosed with Metabolic Associated Steatotic Liver Disease (MASLD), or people who have been identified as being at risk for developing MASH
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2025-12-23 (Estimated)

PRIMARY OUTCOMES:
Description of awareness, understanding, and perception of MASLD/MASH, comorbidities, and risk factors | At the time of survey (Day 1)
  Healthcare Provider (HCP) Quantitative Segment 7-point Likert scale
  1 indicates very strongly disagree and 7 indicates very strongly agree
Description of awareness, understanding, and perception of MASLD/MASH, comorbidities, and risk factors | At the time of survey (Day 1)
  Patient Quantitative Segment 7-point Likert scale
  1 indicates very strongly disagree and 7 indicates very strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (5):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Puteaux, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com